CLINICAL TRIAL: NCT06053138
Title: Assessment of BHB Concentration Agreement Among Sampling Locations and the Impact of Ketosis on Erythropoietin Levels: A Two-Part Study
Brief Title: Assessment of BHB Concentration Agreement Among Sampling Locations and the Impact of Ketosis on EPO, and More
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1-16-02-279-23
Record Dates: First submitted 2023-08-23; First posted 2023-09-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2023-08

CONDITIONS: Ketosis
Keywords: ketosis; ketone monoester; erythropoitin; sex hormones
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: Participants are all exposed to the intervention (ketosis) in part 1 followed by randomization to either active intervention (ketosis) or placebo in part 2 of the study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants are blinded to the drink (intervention) being either ketosis (obtained by ingestion of a ketone monoester drink) or plaacebo (a tate and volume matched drink). Drinks are provided in similar neutral unlabelled bottles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketosis (Experimental): Ketosis (the condition being investigated) is obtained by ingestion of a ketone monoester
  Interventions: Dietary Supplement: Ketone monoester
- Control (Placebo Comparator): The control arm is a drink matched in taste, volume, appearence, and viscosity to that of the active/experimental arm
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone monoester — Supraphysiological levels of ketosis acutely, part 1, and intermittently and longer lasting, part 2, as obtained by ingestion of a ketone monoester dietary supplement
  Other Names: KetoneAid Ke4 Pro Ketone Ester
  Arms: Ketosis
Dietary Supplement: Placebo — The placebo vehicle is matched to the ketosis intervention in the experimental arm with regards to taste, volume, viscosity, appearence, and packaging
  Arms: Control

SUMMARY:
his study aims to address two key aspects - part 1: the suitability of selecting a specific sampling site for BHB measurement in patients and research, as well as potential differences between capillary and venous blood measurements.

Additionally, the study will delve into the effects of ketosis on EPO concentrations, sex hormones levels, and hemodynamic markers and blood pressure - part 2. This investigation will utilize blood samples collected during part 1, including acute effects, as well as samples taken on day 7 and day 14 during which period participants are exposed to intermittent ketosis.

DETAILED DESCRIPTION:
Aim and Perspective:

The primary objective of this study - part 1 - is to ascertain:

The agreement between estimates of beta-hydroxybutyrate (BHB) in capillary and venous blood and whether this agreement is influenced by the level of BHB.

The agreement in BHB measurements between finger and earlobe capillary samples. The agreement in BHB measurements between venous estimates obtained through a point-of-care device (KetoSure) and full blood estimates obtained through hydrophilic interaction liquid chromatography tandem mass spectrometry (HLCMS).

The central aim of the study - part 2 - is to investigate:

The impact of ketosis on short-term and long-term erythropoietin (EPO) levels. The resulting effects of EPO on erythropoiesis and iron metabolism during a two-week period of intermittent ketosis.

The effects of ketosis and sex hormones including derived factors The effects of ketosis on hemodynamic markers and blood pressure

The study aims to determine the appropriateness of selecting a specific sampling site for BHB measurement in both patient care and research. Additionally, it seeks to identify any differences between BHB measurements from capillary and venous blood samples. The study will also examine the concordance between the KetoSure point-of-care-test (POCT) device and the established gold standard, offering insight into any discrepancies arising from electrochemical estimations and HLCMS. Accurate BHB measurement is crucial in clinical and experimental settings. Firstly, precise BHB quantification can inform clinical decision-making for conditions such as suspected hyperinsulinemia, uncertain etiology hypoglycemia, and diabetic ketoacidosis. Secondly, given the extensive research on BHB inference and ketones in recent years, the credibility of these studies heavily hinges on the precision of measurements concerning sample type and sampling site selection.

Additionally, during part 2 of the study, the effects of ketosis on EPO concentrations, sex hormone levels, hemodynamic markers, and blood pressure measurements will be explored. These analyses will be conducted using blood samples collected during part 1 (acute effects) as well as on day 7 and day 14, when participants experience intermittent ketosis.

Analytical Approach:

Following a visual assessment of graphical linearity representation, differences will be calculated using the paired t-test, agreement determined using the Bland-Altman plot, and correlations assessed using Pearson's r. Further calculations will employ Lin's concordance correlation coefficient of absolute agreement. For comparisons across observations in parts 1 and 2, an analysis equivalent to repeated measurements ANOVA will be applied. No imputation of missing data will be conducted, and steps will be taken to ensure data completeness before participants leave the research facilities.

Sample Size and Power Calculation:

Given the absence of prior studies on BHB agreement data, our study's sample size calculations are based on relevant literature. Citing Boyd et al., and considering correlated glucose estimates, a sample size of 13 participants will provide sufficient statistical power (alpha = 0.05, beta = 20%) to detect a difference of 0.58 mM in glucose estimates between capillary and venous blood samples (SD = 0.68 mM). A sample size of 20 participants is justifiably required to detect a clinically significant difference of 1 mM (SD = 1.5) under the same parameters. Consequently, we will include 16 patients in our study, aligning with similar projects and justified sample size for part 2.

Collection of New Biological Material:

A total of 150 mL of blood will be drawn, including incidental spillage from repeated sampling through an indwelling catheter in part 1. No spillage is expected in part 2 as blood sampling occurs only twice in an outpatient setting, with subsequent laboratory analysis.

Purpose of Storage:

All biological samples will be stored for the entire data collection period and 18 months thereafter for bulk analysis. Storage will be at -80 ºC. A research biobank will be established to analyze samples not analyzed on the study day, with surplus material preserved for future research.

Handling of Patient Information:

Access to participants' electronic patient records, limited to the laboratory results section, is included in the consent for practical reasons. Only routinely obtained treatment-related information necessary for analysis will be accessed. Any information obtained before consent will be shared with the investigator.

Data Privacy and Sharing:

Data will be pseudonymized during analysis, with de-identification codes retained by the primary investigator. Data access will be restricted to investigators until final analysis. Upon anonymization, other investigators will gain access. After publication, all data will be open accesible upon reasonably request. However, consideration to make data available to public scrutiny is under consideration.

Financial Information:

The study is initiated and financed by the primary investigator, Henrik Holm Thomsen. Funding originates from independent research funds within the Department of Internal Medicine, Regional Hospital Viborg. Additional external funding will be pursued for study expenses only, excluding investigator salaries. Financial transactions follow the research practices of the Central Denmark Region and Regional Hospital Viborg. Research investigators and collaborators have no financial interests in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* BMI 19-30 kg/m2
* Expected ease of catheter insertion
* Considered of sound health
* Oral and written informed consent

Exclusion Criteria:

* Inability to fully understand the consent including consent forms
* Inability to cooperate to the study
* electrolyte disorders
* acute or chronic kidney disease or ompromised renal function including excess risk
* servere hypertension
* autoimmune disease
* liver or bile disease
* diabetes mellitus
* reactive hypoglycemia or similar disorders
* treatment with drugs, and dietary supplements with inference on key metabolic or hormonal markers, e.g. insulin, glucagon, DDP-IV inhibitors, GLP-1 RA, sulfunylurea
* use of illegal or otherwise use of medicinal products without prescription
* anemia or other know disease of the hematopoietic system
* previous bariatric surgery
* previous myocardial infarction or uncontrolled myocardial ischemia
* recent intended/unintended weight loss
* allergies to catheters or adhesives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Plasma Beta-hydroxybutyrate (BHB) | Baseline (0 minutes), 30, 60, 90, 120, 150, and 180 minutes(part 1) and at Day 8 and Day 15 (part 2)
  The levels of BHB were measured using the Ketosure POCT device, with samples taken from capillary blood (finger pulp and earlobes) and venous plasma. Plasma-BHB was also measured using LCMS on venous blood samples. Measured and reported in mmol/L (millimoles per liter)
Erythropoietin (EPO) | Baseline (0 minutes),60, 90, 150, and 180 minutes(part 1) and at Day 8 and Day 15 (part 2)
  EPO concentrations measured in blood samples on standard hospital laboratory equipment. Measured and reported in IU/L (international units per liter)
Testosterone | Baseline (0 minutes), 90, and 180 minutes(part 1) and at Day 8 and Day 15 (part 2)
  Measured in venous plasma. Measured and reported in nmol/L (nanomoles per liter) pmol/L (picomoles per liter) for estradiol
Aldosterone | Baseline (0 minutes), 90, and 180 minutes (part 1) and at Day 8 and Day 15 (part 2)
  Hemodynmiac and blood pressure regulating hormones measured in plasma. Measured and reported in standard units: pmol/L (picomoles per liter), renin in mIU/L (milli international units per liter), proBNP in ng/L (nanogram per liter)
Estradiol | Baseline (0 minutes), 90, and 180 minutes (part 1) and at Day 8 and Day 15 (part 2)
  Measured in pmol/L (picomoles per liter) in venous plasma
Renin | Baseline (0 minutes), 90, and 180 minutes (part 1) and at Day 8 and Day 15 (part 2)
  Venous plasma, reported in mIU/L (milli international units per liter)
ProBNP | Baseline (0 minutes), 90, and 180 minutes (part 1) and at Day 8 and Day 15 (part 2)
  Measured in venous plasma and reported in ng/L (nanogram per liter). proBNP=pro brain natriuretic peptide

OTHER OUTCOMES:
Hematocrit | Baseline (0 minutes), 90, and 180 minutes(part 1) and at Day 8 and Day 15 (part 2)
  hematocrit - percentages
  mean corpuscular volume - fmol (femtomoles) ferritin - microgram/L transferrin - microgram/L
  Measured and reported in standard units
Hemoglobin | Baseline (0 minutes), 90, and 180 minutes(part 1) and at Day 8 and Day 15 (part 2)
  hemoglobin - mmol/L hematocrit - percentages hemoglobin - mmol/L erythrocytes - x10^12/L leukocytes - x10^12/L mean corpuscular volume - fmol (femtomoles) ferritin - microgram/L transferrin - microgram/L
  Measured and reported in standard units
Erythrocytes | Baseline (0 minutes), 90, and 180 minutes(part 1) and at Day 8 and Day 15 (part 2)
  erythrocytes - x10^12/L hematocrit - percentages hemoglobin - mmol/L erythrocytes - x10^12/L leukocytes - x10^12/L mean corpuscular volume - fmol (femtomoles) ferritin - microgram/L transferrin - microgram/L
  Measured and reported in standard units
Leukocytes | Baseline (0 minutes), 90, and 180 minutes(part 1) and at Day 8 and Day 15 (part 2)
  leukocytes - x10^12/L hematocrit - percentages hemoglobin - mmol/L erythrocytes - x10^12/L leukocytes - x10^12/L mean corpuscular volume - fmol (femtomoles) ferritin - microgram/L transferrin - microgram/L
  Measured and reported in standard units
Mean corpuscular volume | Baseline (0 minutes), 90, and 180 minutes(part 1) and at Day 8 and Day 15 (part 2)
  mean corpuscular volume - fmol (femtomoles) hematocrit - percentages hemoglobin - mmol/L erythrocytes - x10^12/L leukocytes - x10^12/L mean corpuscular volume - fmol (femtomoles) ferritin - microgram/L transferrin - microgram/L
  Measured and reported in standard units
Lutropin | Baseline (0 minutes), 90, and 180 minutes(part 1) and at Day 8 and Day 15 (part 2)
  lutropin - IU/L (international units per liter)
Follitropin | Baseline (0 minutes), 90, and 180 minutes(part 1) and at Day 8 and Day 15 (part 2)
  follitropin - IU/L
Home blood pressure measurements | Measurements are made just prior to Day 8 and Day 15 in addition to measurements in Study part 1 made by research staff
  Study participants record their home blood pressure and heart rate, both systolic and diastolic, with provided automated blod pressure measurement devices in accordance with guidelines. Blood pressure is estimated and reported in mmHg
Heart rate | Measurements are made just prior to Day 8 and Day 15 in addition to measurements in Study part 1 made by research staff
  heart rate measured in beats per minut with the blood pressure monitor that also counts the heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Henrik H Thomsen, Ph.D., Principal Investigator — Department of Internal Medicine, Viborg Regional Hospital, Denmark
Locations (1):
- Department of Internal Medicine, Viborg Regional Hospital, Viborg, Denmark

IPD SHARING:
Plan to Share IPD: No